CLINICAL TRIAL: NCT04027725
Title: Pilot Study Evaluating the Effectiveness of Neurofeedback Training in the Improvement of Cognitive Functions of the Elderly With Mild Cognitive Impairment
Brief Title: NEUROFEEDBACK TRAINING FOR OLDER ADULTS WITH MILD COGNITIVE IMPAIRMENT: A PILOT STUDY
Acronym: NEUROFEEDEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K170908J; 2017-A02933-50 (Other: ID-RCB (ANSM))
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive Impairment; Neurofeedback; Electroencephalography; Memory; Attention
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor neurofeedback training group (Experimental): Three interventions will be administered :
  * An electroencephalography recording (EEG) for 30 minutes with an electrocap of 19 scalp locations according to the international 10-20 EEG placement system.
  * The second intervention is the neuropsychological assessments and questionnaires. They will be done in one session for approximately 2hours.
  * The third intervention is the neurofeedback training sensorimotor that will be recorded at channel Cz according to the international 10-20 system.
  Interventions: Behavioral: Neurofeedback
- Control Group (No Intervention): Three interventions will be administered :
  * An electroencephalography recording (EEG) for 30 minutes with an electrocap of 19 scalp locations according to the international 10-20 EEG placement system.
  * The second intervention is the neuropsychological assessments and questionnaires. They will be done in one session for approximately 2hours
  * The psychopedagogical care: each session will be organized using the same video material

INTERVENTIONS:
Behavioral: Neurofeedback — Neurofeedback experiment will consist of 20 sessions of neurofeedback training, twice or three times a week during seven weeks. Each session will last for 40 minutes. The experimental group will undergo questionnaires, EEG recording and neuropsychological assessments in three-time points, pre-training (T0), post-trianing (T1) and 1 month follow-up (T2). Electroencephalography will be recorded by a technician in EEG for each participant, EEG power spectrum will be calculated in pre (T0) and post neurofeedback training/psycho-pedagogical care at T1 and T2.
  Other Names: Electroencephalography
  Arms: Sensorimotor neurofeedback training group

SUMMARY:
The purpose of this study is to evaluate the effects of SMR neurofeedback training on cognitive performance and electrical brain activity in elderly with cognitive impairment.

DETAILED DESCRIPTION:
Older adults with Mild Cognitive Impairment (MCI) are at high risk to progress to Alzheimer's disease (AD). Slowing down effect of dementia by enhancing brain plasticity represents on of the most prominent challenges. Neurofeedback is one of the promising techniques that showed therapeutic efficacy and cognitive improvement in attention-deficit hyperactivity disorder, epilepsy, stroke. The investigators aim to study the effects of a sensorimotor neurofeedback training protocol (SMR) on cognitive performances in elderly and to assess whether MCI patients change in brain electrical activity after training.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Mild Cognitive Impairment, educational level of 9 years of studies minimum, righthandedness, subjective memory complaint confirmed by an informant, a mini mental Status Examination score > 20, preserve activity of daily living and absence of dementia.

Exclusion Criteria:

Elderly persons who were under guardianship, resident in nursing facilities, neurological disease, psychiatric disease and involved in another cognitive intervention.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change on Rey Auditory Verbal Learning test | Baseline assessment in 2 weeks period before intervention, change from baseline at immediately after the end of the intervention , and after 1-month follow-up
  Assessment of Verbal learning in episodic memory

SECONDARY OUTCOMES:
relative power for delta, theta, alpha, sensorimotor and lower beta frequency bands. | assessment at baseline, change from baseline to immediately after the NF training and 1 month follow-up
  Description : Electroencephalography was recorded and EEG power spectrum was calculated using the fast Fourier Transform. The power spectral density was calculated to extract the relative power for each frequency band and estimated as a log-ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie RIGAUD, Professor, Principal Investigator — APHP
Locations (1):
- Hopital BROCA, Paris, France

IPD SHARING:
Plan to Share IPD: No